CLINICAL TRIAL: NCT05677178
Title: Response Prediction in EBV-HLH Using Metabonomics Analysis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Head of the hematology department, Beijing Friendship Hospital
Other Study IDs: 2022-P2-092-01
Record Dates: First submitted 2022-11-10; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-11

CONDITIONS: Hemophagocytic Lymphohistiocytoses; EBV; Metabonomics
Keywords: Hemophagocytic Lymphohistiocytoses; EBV; matabonomics
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- survival group: Patients who survived 2 months after treatment.
  Interventions: Other: observational
- death group: Patients who died 2 months after treatment.
  Interventions: Other: observational

INTERVENTIONS:
Other: observational — This study is an observational study without any intervention.

SUMMARY:
Hemophagocytic lymphohistiocytosis (HLH) is a rare, poorly recognized and underdiagnosed syndrome of excessive immune activation, which is rapidly fatal. Epstein-Barr virus (EBV) is a common trigger of HLH, particularly in Asian individuals. We aim to analyze metabolomics and cytokine profiles of patients before and after treatment to explore the metabolomic characteristics of EBV-HLH, and search for pathogenic mechanisms and therapeutic targets.

DETAILED DESCRIPTION:
Hemophagocytic lymphohistiocytosis (HLH) is a rare, poorly recognized and underdiagnosed syndrome of excessive immune activation, which is rapidly fatal. Without early intervention, the median survival time is less than 2 months.Epstein-Barr virus (EBV) is a common trigger of HLH, particularly in Asian individuals. We aim to analyze metabolomics and cytokine profiles of patients before and after treatment to explore the metabolomic characteristics of EBV-HLH, and search for pathogenic mechanisms and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet HLH-04 diagnostic criteria
* EBV-DNA viral load in the peripheral blood > 500 copies/mL
* Informed consent obtained.

Exclusion Criteria:

* refuse to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who were diagnosed with EBV-HLH in China.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Difference in metabonomics pattern between subgroups | 2 months
  Compare metabonomics pattern of the survival group with that of the death group, identify potential predictors of outcomes, and establish a survival prediction model in patients with EBV-HLH. Measure metabolite levels.
Difference in cytokine pattern between subgroups | 2 months
  Compare metabonomics and cytokine pattern of the survival group with that of the death group, identify potential predictors of outcomes, and establish a survival prediction model in patients with EBV-HLH. Measure cytokine levels.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No